CLINICAL TRIAL: NCT06996262
Title: The Relationship Between NOVA-Classified Processed Food Intake and Cardiometabolic Risk Factors in Türkiye
Brief Title: Cardiometabolic Risk Factors and Processed Food
Status: Completed | Type: Observational
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Hande Seven Avuk, Assistant Professor, Head of Nutrition and Dietetic Department, Istanbul Bilgi University
Other Study IDs: ULTRAHEARTTR
Record Dates: First submitted 2025-05-19; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Disease; Cardiovascular Diseases; Nutrition; Nutritional Disease; Cardiometabolic Diseases; Cardiometabolic Risk Factors
Keywords: processed food; cardiometabolic risk; obesity; Framingham risk score
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Nutrition Disorders; Obesity | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Study Group: * Aged 18-65,
  * Volunteers at the Zonguldak Atatürk State Hospital
  * Outpatients applying to the internal medicine polyclinic
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — The questionnaire consisted of structured questions covering sociodemographic information, health status, dietary habits, and physical activity levels.
Other: observational study — Anthropometric measurements was taken.
Other: observational study — Biochemical analyses were measured was measured using routine methods.
Other: observational study — Blood pressure were measured was measured using routine methods.

SUMMARY:
Cardiovascular diseases (CVD) remain a primary cause of chronic disability and mortality globally, with cardiometabolic risk factors such as hypertension, dyslipidemia, obesity, and diabetes significantly contributing to their development. Poor nutrition is recognized as a modifiable key risk factor for CVD, representing a crucial area for prevention strategies. While current research often emphasizes overall dietary patterns and quality in CVD prevention, the spectrum of food processing, ranging from minimally processed to ultra-processed foods (UPFs), can profoundly influence diet quality.

Ultra-processed foods, characterized by industrial processing techniques, additives, and special industrial ingredients, have been shown to potentially compromise the health benefits of food by reducing essential nutrients and bioactive compounds, introducing unhealthy elements, and altering food structures. Emerging epidemiological evidence links higher UPF consumption to an increased risk of obesity, hypertension, metabolic syndrome, and type 2 diabetes, with studies like the Framingham Offspring Study indicating a positive association with CVD incidence.

Globally, UPF consumption is on the rise, constituting a significant portion of daily energy intake. In Turkey, data from the 2021 National Nutrition and Health Survey reveals that a substantial 58% of adults consume processed foods daily . This is particularly concerning given Turkey's high burden of CVD, which has been the leading cause of mortality for decades and is projected to increase further due to an aging population and rising rates of diabetes and obesity. Notably, Turkey has the highest rate of early myocardial infarction in Europe.

Given the increasing consumption of UPFs and their potential health implications, especially in a country with a high prevalence of CVD like Turkey, understanding the relationship between dietary factors and cardiovascular health is critical. Therefore, this study aims to investigate the association between processed food intake and cardiometabolic risk factors among adult individuals in Türkiye.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years
* volunteers patients

Exclusion Criteria:

* people under 18 years of ages
* people over 65 years of ages
* pregnant and breastfeeding women
* individuals with active cancer or chronic illnesses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients applying to the internal medicine polyclinic
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Biochemical Measurements - Fasting blood glucose | Baseline
  Fasting blood sugar (mg/dL) will be analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse.
Biochemical Measurement - Lipid Profile | Baseline
  Participants' biochemical tests (total cholesterol, HDL cholesterol, LDL cholesterol, triglyceride, (mg/dL) were analyzed in the hospital biochemistry laboratory using routine methods at the beginning of the study from blood samples taken by a nurse after at least 12 hours of fasting and without consuming alcohol for 24 hours before.
Biochemical Measurements - HbA1C | Baseline
  Fasting blood sugar (mg/dL) was analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse at the beginning of the study.
Biochemical Measurements - Uric acid | Baseline
  Participants' serum uric acid tests (mg/dL) was analyzed in the hospital biochemistry laboratory using routine methods at the beginning of the study from blood samples taken by a nurse after at least 12 hours of fasting and without consuming alcohol for 24 hours before.
Blood Pressures | Baseline
  Systolic and Diastolic blood pressure (mmHg) includes auscultation of the brachial artery with a stethoscope to detect the appearance and muffled or absent Korotkoff sounds.
Framingham Risk Score | Baseline
  The Framingham Risk Score was used to assess the risk of cardiovascular disease (CVD) in participants. To evaluate the 10-year risk of cardiovascular events, the following variables were considered: age, gender, total cholesterol, HDL cholesterol, systolic and diastolic blood pressure, smoking status, and diabetes. Each variable is assigned a specific score, and the total score for each participant is calculated by summing these. A higher score indicates a greater cardiometabolic risk.
Framingham Risk Percentage | Baseline
  The total Framinham risk score estimates the probability of experiencing a cardiovascular event within 10 years, and the resulting percentage values are classified into low, moderate, and high risk categories.
  * Low risk: Individuals with a score of less than 10%. This suggests a relatively low likelihood of experiencing a cardiovascular event within 10 years.
  * Moderate risk: Individuals with a score between 10% and 20%.
  * High risk: Individuals with a score above 20%.
Anthropometric Measurements - Body weight (kg) | Baseline
  At the beginning of the study, body weights (kg) was measured using a calibrated portable digital scale with a sensitivity of 50 grams in accordance with the measurement standards.
Anthropometric Measurements - Height | Baseline
  Height (cm) was measured with a stadiometer in the Frankfort plane, standing and with the head upright.
Body Mass Index | Baseline
  The body mass index (BMI) of the participants was calculated according to the body weight (kg) / height (m)2 formula.
Body Mass Index Classification | Baseline
  The body mass index (BMI) of the participants is classified according to the World Health Organization (WHO) criteria. BMI ≤ 18.5 kg/m2 is underweight, between 18.5-24.99 kg/m2 is normal, ≥ 25 kg/m2 is overweight, and ≥ 30 kg/m2 is obese.
Anthropometric Measurements - Waist circumference | Baseline
  The waist circumference was measured with a non-flexible tape measure at the midpoint between the lowest rib and the crystalline prominence.
Anthropometric Measurements - Hip circumference | Baseline
  The individual was asked to stand upright with their arms at their sides and their feet side by side when measuring hip circumference. The Frankfort plane was provided. The individual was measured with a tape measure from the right side, determining the highest point of the hip (from the side).
Anthropometric Measurements - Waist/Hip Ratio | Baseline
  Waist/hip ratio was obtained by dividing waist circumference by hip circumference.
Anthropometric Measurements - Waist/Height Ratio | Baseline
  Waist/height ratio was obtained by dividing waist circumference by height.
Anthropometric Measurements - Neck Circumference | Baseline
  Neck circumference (cm) was measured at the level of the laryngeal prominence using a flexible tape measure, with participants standing, their heads upright and their eyes looking straight ahead.
Food Frequency Record | Baseline
  Food frequency records were taken to assess processed and ultra-processed food consumption according to the Nova classification.

SECONDARY OUTCOMES:
Physical Activity Levels | Baseline
  The International Physical Activity Questionnaire (IPAQ) Short Form, developed by Craig et al. and whose Turkish validity and reliability study was conducted by Öztürk, were used to assess the physical activity levels of the participants. In the IPAQ short form (7 questions) assessment, the energy required for activities will be calculated with the Metabolic Equivalent Task minutes per week (MET-minutes) score. The calculation of the total score includes the sum of the duration (minutes) and frequency (days) of walking, moderate-intensity activity and vigorous activity.
Physical Activity Levels Classification | Baseline
  Physical activity will be classified into 3 groups according to MET value. The physically inactive group is determined as those below 600 MET-min/week, moderately active between 600-3000 MET-min/week, active above 3000 MET-min/week, very active above 1500 MET-min/week and at least 3 days of vigorous activity or above 3000 MET-min/week and at least 7 days of walking.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Seven Avuk, PhD, Principal Investigator — Istanbul Bilgi University
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tokgozoglu L, Kayikcioglu M, Ekinci B. The landscape of preventive cardiology in Turkey: Challenges and successes. Am J Prev Cardiol. 2021 Apr 14;6:100184. doi: 10.1016/j.ajpc.2021.100184. eCollection 2021 Jun. PMID 34327504
- [Background] Hosseininasab D, Shiraseb F, Noori S, Jamili S, Mazaheri-Eftekhar F, Dehghan M, da Silva A, Bressan J, Mirzaei K. The relationship between ultra-processed food intake and cardiometabolic risk factors in overweight and obese women: A cross-sectional study. Front Nutr. 2022 Aug 9;9:945591. doi: 10.3389/fnut.2022.945591. eCollection 2022. PMID 36017229
- [Background] Elizabeth L, Machado P, Zinocker M, Baker P, Lawrence M. Ultra-Processed Foods and Health Outcomes: A Narrative Review. Nutrients. 2020 Jun 30;12(7):1955. doi: 10.3390/nu12071955. PMID 32630022
- [Background] Juul F, Martinez-Steele E, Parekh N, Monteiro CA, Chang VW. Ultra-processed food consumption and excess weight among US adults. Br J Nutr. 2018 Jul;120(1):90-100. doi: 10.1017/S0007114518001046. Epub 2018 May 6. PMID 29729673
- [Background] Monteiro CA, Cannon G, Levy RB, Moubarac JC, Louzada ML, Rauber F, Khandpur N, Cediel G, Neri D, Martinez-Steele E, Baraldi LG, Jaime PC. Ultra-processed foods: what they are and how to identify them. Public Health Nutr. 2019 Apr;22(5):936-941. doi: 10.1017/S1368980018003762. Epub 2019 Feb 12. PMID 30744710
- [Background] Juul F, Vaidean G, Parekh N. Ultra-processed Foods and Cardiovascular Diseases: Potential Mechanisms of Action. Adv Nutr. 2021 Oct 1;12(5):1673-1680. doi: 10.1093/advances/nmab049. PMID 33942057
- [Background] Juul F, Vaidean G, Lin Y, Deierlein AL, Parekh N. Ultra-Processed Foods and Incident Cardiovascular Disease in the Framingham Offspring Study. J Am Coll Cardiol. 2021 Mar 30;77(12):1520-1531. doi: 10.1016/j.jacc.2021.01.047. PMID 33766258
- [Derived] Ozkan I, Ozlu Karahan T, Seven Avuk H. Processed Food Consumption Based on the NOVA Classification Is Associated With Elevated Cardiometabolic Risk in Turkish Adults. Food Sci Nutr. 2025 Sep 26;13(10):e71014. doi: 10.1002/fsn3.71014. eCollection 2025 Oct. PMID 41019184
- See also: Ministry of Health, General Directorate of Public Health. (2022). Türkiye Nutrition Guide (TUBER) 2022. Ministry of Health Publication No: 1031. Ankara: Ministry of Health. — https://hsgm.saglik.gov.tr/depo/birimler/saglikli-beslenme-ve-hareketli-hayat-db/Dokumanlar/Rehberler/Turkiye_Beslenme_Rehber_TUBER_2022_min.pdf